CLINICAL TRIAL: NCT06631417
Title: A Trial to Investigate Relative Bioavailability of Three Different BI 1291583 Formulations Following Oral Administration at Two Dose Levels to Healthy Subjects (an Open-label, Randomised, Single-dose, Three-period Crossover Trial Consisting of 2 Parts)
Brief Title: A Study in Healthy People to Test How 2 Different Doses of BI 1291583 Are Taken up in the Body When Given in 3 Different Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0021; 2023-510260-13-00 (Registry Identifier: CTIS); U1111-1301-1371 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Study has 2 parts, participants cross over between 3 treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1291583 formulation 1 then formulation 2 then formulation 3 (part A) (Experimental)
  Interventions: Drug: BI 1291583
- BI 1291583 formulation 1 then formulation 2 then formulation 3 (part B) (Experimental)
  Interventions: Drug: BI 1291583

INTERVENTIONS:
Drug: BI 1291583 — formulation 1
  Other Names: Verducatib
Drug: BI 1291583 — formulation 2
  Other Names: Verducatib
Drug: BI 1291583 — formulation 3
  Other Names: Verducatib

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of two different formulations of BI 1291583 (test formulations) compared to BI 1291583 reference formulation administered at two different dose levels.

ELIGIBILITY:
Inclusion Criteria :

1. Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. For female subjects: a subject who meets any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 5 months after the last trial medication administration:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
   * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
   * Sexually abstinent
   * A vasectomized sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial subject
   * Surgically sterilised (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal occlusion)
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria :

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | Up to 22 days
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 22 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞) | Up to 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com